CLINICAL TRIAL: NCT03982693
Title: Trial to Assess Chelation Therapy in Critical Limb Ischemia
Acronym: TACT3a
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mt. Sinai Medical Center, Miami (Other)
Responsible Party: Principal Investigator, Gervasio Lamas, MD, Principal Investigator, Mt. Sinai Medical Center, Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-05-H-01
Record Dates: First submitted 2019-05-27; First posted 2019-06-11 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Critical Limb Ischemia; Diabetes
Keywords: Chelation; Critical Limb Ischemia; Diabetes
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Diabetes Mellitus | interventions — Pentetic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): edetate disodium (EDTA)dff active infusion
  Interventions: Drug: Edetate Disodium
- Placebo (Placebo Comparator): Placebo infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Edetate Disodium — The solution contains up to 3 g of edetate disodium adjusted based on creatinine clearance, 2 g of magnesium chloride, 100 mg of procaine hydrochloride, 2500 U of heparin, 7 g of ascorbate, 2 milliequivalent (mEq) potassium chloride (KCl), 840 mg sodium bicarbonate, 250 mg pantothenic acid, 100 mg of thiamine, 100 mg of pyridoxine, and sterile water to complete 500 mL.
  Other Names: TACT EDTA infusion
  Arms: Active
Other: Placebo — Placebo infusions consist of 500 ml normal saline.
  Arms: Placebo

SUMMARY:
TACT3a is a double blind, placebo-controlled, randomized trial to test a novel therapy, edetate disodium-based chelation of environmentally acquired toxic metals, to reduce cardiovascular events including amputation in high-risk diabetic patients.

DETAILED DESCRIPTION:
TACT3a is a double blind, placebo-controlled, randomized trial to test a novel therapy, edetate disodium-based chelation of environmentally acquired toxic metals, to reduce cardiovascular events including amputation in high-risk diabetic patients.

The study plans to enroll 50 patients with diabetes and critical limb ischemia (CLI) to prevent the major cardiovascular endpoints of major amputation, coronary revascularization, stroke, Myocardial Infarction (MI), or death (all-cause) during an average 1.25 years of follow-up. Patients will be randomly assigned to chelation or placebo with a 3:2 (30 active, 20 placebo) allocation ratio. Treatment will consist of 40 active or placebo infusions over 30 weeks. Active therapy will be the same edetate disodium-based infusion used safely and successfully in a previous published study, Trial to Assess Chelation Therapy (TACT). Baseline and post infusion urine metals will be collected. Following the final infusion, patients will be contacted quarterly until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* History of diabetes, defined as medical record evidence or patient report of currently using insulin or oral hypoglycemic agents, or with a history of fasting blood glucose measurement of 126 mg/dL or higher, or a history of HbA1c of 6.5% or higher.
* Significant stenosis (≥ 75%) of two or more infra-popliteal arteries in the affected limb as verified by at least one imaging technique (angiography, magnetic resonance angiogram, coronary computed tomography angiogram, or doppler examination) within 6 months prior to enrollment;
* History of CLI defined as moderate or high-risk infra-popliteal chronic critical limb ischemia (Rutherford Clinical Severity Score 4 or 5) defined as:

  * The presence of rest pain or non-healing ulceration or gangrene for at least 2 weeks plus documentation of severely compromised tissue perfusion:
  * If there is tissue loss, a resting ankle systolic pressure of ≤ 60 mmHg in the affected limb; or a resting toe systolic pressure of ≤ 40 mmHg or a tissue perfusion pressure (TPP) <40 mmHg.
  * If there is no tissue loss, a resting ankle pressure of ≤ 50 mmHg or resting toe systolic pressure of ≤ 30 mmHg or a tissue perfusion pressure (TPP) < 30 mmHg.
* Not a candidate or a failed candidate for surgical or transcatheter revascularization;
* Able to give informed consent.

Exclusion Criteria:

* <7 days following lower extremity (infra-popliteal), carotid, or coronary revascularization.
* Arterial insufficiency in the lower extremity as the result of a non-atherosclerotic disorder.
* Subjects with evidence of active infection (e.g., cellulitis, osteomyelitis) or deep ulceration exposing bone or tendon or extensive heel ulceration
* Subjects with extensive gangrene extending above the MT joint
* Subjects in whom there is severe pain at rest uncontrollable with pain medications
* Prior intravenous chelation therapy consisting of > 1 infusion within 5 years; if only 1 infusion took place, patient cannot be enrolled for at least 12 months after said infusion.
* Oral chelation with an FDA-approved chelating agent within 2 years
* Allergy to any components of the study drug
* Planned leg revascularization within 1 month of enrollment
* Symptomatic or clinically evident acute heart failure
* Heart failure hospitalization within 3 months
* Blood pressure >160/100
* No venous access
* eGFR < 30 mL/min per 1.73 m2 or lower (CKD stages 1-3) calculated with MDRD
* Known or suspected acute kidney injury using prevalent KDIGO criteria45
* Platelet count <100,000/mm3
* Cigarette smoking within the last 3 months
* Liver disease or Alanine aminotransferase (ALT), aspartate aminotransferase (AST) > 2.0 times the upper limit of normal (this will require clearance by the Study PI)
* Diseases of copper, iron, or calcium metabolism (other than osteopenia or osteoporosis, or simple iron deficiency). These require evaluation by the Study PI
* Inability to tolerate the study-required fluid load
* Other medical condition likely to affect patient survival within 3 years
* Women of child-bearing potential
* Any factor that suggests that the potential participant will not be able to adhere to the protocol.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Prevention of major cardiovascular endpoints | 3 years (average follow-up 1.25 years)
  Major cardiovascular endpoints include: coronary revascularization, stroke, MI, death (all-cause), or major amputation

SECONDARY OUTCOMES:
Amputations | 3 years (average follow-up 1.25 years)
  * Major amputations due to vascular disease. Major amputations are defined as any procedure that results in amputation at the level above the ankle. 49, 50
  * Total amputations due to vascular disease
Heart failure | 3 years (average follow-up 1.25 years)
  • Heart failure hospitalizations or prolonged (>12 hours) ER stay for heart failure
Changes in Pain severity | 3 years (average follow-up 1.25 years)
  • Any changes in pain will be recorded at baseline, infusions 10, 20, 40 (or final), and end of study recorded using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference- Short Form 8a. The scale range is 1 to 5, with 1 being the best outcome (no pain interference) and 5 the worse (very much interference)
Urine Metals | 1 year
  • Changes in urine metal levels measured at the Metals Core Lab and measured at baseline and infusion 40 (or final).
Changes in Quality of Life | 3 years (average follow-up 1.25 years)
  • Health-related quality of life (QOL) changes recorded at baseline, 10, 20, 40 (or final), and end of study using the 36-Item Short Form Health Survey (SF-36 v2). The 36 questions assess eight health-related concepts: physical functioning, role limitations due to physical health problems (role physical), bodily pain, general health, energy levels/fatigue (vitality), social functioning, role limitations due to emotional problems (role emotional), and psychological distress (mental health). The scales vary depending on the question asked.The survey will be used to detect change (better or worse) in participants' health state over the course of the study.
Wound Severity | 3 years (average follow-up 1.25 years)
  Wound severity (quantified and imaged with HIPAA-compliant photography) photographed at baseline 10, 20, 40 (or final), and end of study
Changes in skin perfusion pressure in the ankle | 3 years (average follow-up 1.25 years)
  • Changes in skin perfusion pressure will be measured at 10, 20, 40 (or final), and end of study, using the ankle-brachial index (mmHg)
Changes in skin perfusion pressure in the toe | 3 years (average follow-up 1.25 years)
  • Changes in skin perfusion pressure will be measured at 10, 20, 40 (or final), and end of study, using the toe-brachial index (mmHg).
Changes in PAD Quality of Life | 3 years (average follow-up 1.25 years)
  • PAD related quality of life (QOL) changes recorded at baseline, 10, 20, 40 (or final), and end of study using the Peripheral Artery Questionnaire (PAQ), which is a 20-item questionnaire measuring physical limitations, symptoms, symptom stability, treatment satisfaction, quality of life, and social function. The scales vary depending on the question asked. The survey will be used to detect change (better or worse) in participants responses over the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Gervasio Lamas, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, Miami Beach, Florida, United States

REFERENCES:
- [Background] Arenas IA, Navas-Acien A, Ergui I, Lamas GA. Enhanced vasculotoxic metal excretion in post-myocardial infarction patients following a single edetate disodium-based infusion. Environ Res. 2017 Oct;158:443-449. doi: 10.1016/j.envres.2017.06.039. Epub 2017 Jul 6. PMID 28689036
- [Background] Lamas GA, Goertz C, Boineau R, Mark DB, Rozema T, Nahin RL, Drisko JA, Lee KL. Design of the Trial to Assess Chelation Therapy (TACT). Am Heart J. 2012 Jan;163(1):7-12. doi: 10.1016/j.ahj.2011.10.002. PMID 22172430
- [Background] Escolar E, Lamas GA, Mark DB, Boineau R, Goertz C, Rosenberg Y, Nahin RL, Ouyang P, Rozema T, Magaziner A, Nahas R, Lewis EF, Lindblad L, Lee KL. The effect of an EDTA-based chelation regimen on patients with diabetes mellitus and prior myocardial infarction in the Trial to Assess Chelation Therapy (TACT). Circ Cardiovasc Qual Outcomes. 2014 Jan;7(1):15-24. doi: 10.1161/CIRCOUTCOMES.113.000663. Epub 2013 Nov 19. PMID 24254885
- [Background] Ujueta F, Arenas IA, Diaz D, Yates T, Beasley R, Navas-Acien A, Lamas GA. Cadmium level and severity of peripheral artery disease in patients with coronary artery disease. Eur J Prev Cardiol. 2019 Sep;26(13):1456-1458. doi: 10.1177/2047487318796585. Epub 2018 Aug 28. No abstract available. PMID 30152247
- [Background] Ujueta F, Arenas IA, Escolar E, Diaz D, Boineau R, Mark DB, Golden P, Lindblad L, Kim H, Lee KL, Lamas GA. The effect of EDTA-based chelation on patients with diabetes and peripheral artery disease in the Trial to Assess Chelation Therapy (TACT). J Diabetes Complications. 2019 Jul;33(7):490-494. doi: 10.1016/j.jdiacomp.2019.04.005. Epub 2019 Apr 14. PMID 31101487